CLINICAL TRIAL: NCT03181529
Title: Effects of Psilocybin in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00101821
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome measure (GRID-HAMD) will be assessed by raters blinded to randomization condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants will begin psilocybin intervention immediately after study enrollment.
  Interventions: Drug: Psilocybin
- Delayed Treatment (Experimental): Participants will begin the psilocybin intervention 8 weeks after study enrollment.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a moderately high psilocybin dose in the first session and will receive either a moderately high or high psilocybin dose in the second session.

SUMMARY:
The proposed pilot study will assess whether people with major depressive disorder experience psychological and behavioral benefits and/or harms from psilocybin. This study will investigate acute and persisting effects of psilocybin on depressive symptoms and other moods, attitudes, and behaviors. The primary hypothesis is that psilocybin will lead to rapid and sustained antidepressant response, as measured with standard depression rating scales.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 75 years old
* Have given written informed consent
* Have at least a high-school level of education or equivalent (e.g. GED).
* Have a confirmed Diagnostic Statistical Manual (DSM-5) diagnosis of Major Depressive Disorder and currently experiencing a major depressive episode.
* No antidepressant medication for at least 2 weeks (4 weeks for fluoxetine) prior to enrollment.
* Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study.
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine. Participants will be required to be non-smokers.
* Agree not to take any Pro re nata (PRN) medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrilation), prolonged QTc interval (i.e., QTc > 450 msec), artificial heart valve, or Transient Ischemic Attack (TIA) in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including Mono-Amine Oxidase Inhibitors (MAOIs). For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 25% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table

Psychiatric Exclusion Criteria:

* Current antidepressant use
* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Current or history within one year of meeting DSM-5 criteria for a moderate or severe alcohol, tobacco, or other drug use disorder (excluding caffeine)
* Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Has failed to respond to electroconvulsive therapy during the current major depressive episode
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin

Additional Magnetic Resonance Imaging (MRI) Exclusion Criteria:

* Head trauma
* Claustrophobia incompatible with scanning
* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm brain clip
* Inner ear implant
* Prior history as a metal worker and/or certain metallic objects in the body
* History of clinically significant vertigo, seizure disorder, middle ear disorder, or double vision
* Poor vision not adequately corrected (in order to complete emotional processing task)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Levin AW, Lancelotta R, Sepeda ND, Gukasyan N, Nayak S, Wagener TL, Barrett FS, Griffiths RR, Davis AK. The therapeutic alliance between study participants and intervention facilitators is associated with acute effects and clinical outcomes in a psilocybin-assisted therapy trial for major depressive disorder. PLoS One. 2024 Mar 14;19(3):e0300501. doi: 10.1371/journal.pone.0300501. eCollection 2024. PMID 38483940
- [Derived] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target recruitment for this study was 24 study completers. Due to participant drop outs (reasons described in Figure 1 of the study manuscript), we enrolled a total of 27 participants to achieve our target recruitment goals.
Groups:
- Immediate Treatment: Participants will begin psilocybin intervention immediately after study enrollment.
  Psilocybin: Participants will receive a moderately high psilocybin dose in the first session (20 mg/70 kg) and a high dose in the second session (30 mg/70 kg), spaced approximately 1-week apart.
- Delayed Treatment: Participants will begin the psilocybin intervention 8 weeks after study enrollment.
  Psilocybin: Participants will receive a moderately high psilocybin dose in the first session (20 mg/70 kg) and a high dose in the second session (30 mg/70 kg), spaced approximately 1-week apart.
Period: Overall Study
Arm/Group | Immediate Treatment | Delayed Treatment
Started | 15 | 12
Completed | 13 | 11
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Dropped out of study due to sleep difficulties. Sleep difficulties were also reported at screening | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Delayed Treatment | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (13.0) | 35.2 (9.9) | 39.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: The GRID-Hamilton Depression Rating Scale (GRID-HAMD)
Description: The GRID-Hamilton Depression Rating Scale is a 17-item clinician-administered rating scale designed to assess severity of depressive symptoms. The score range for the GRID-HAMD is 0 to 52, with higher score indicating more severe depression. For this clinician-rated measure, a clinically significant response was defined as ⩾50% decrease in measure relative to Baseline; symptom remission was defined as ⩾50% decrease in measure relative to Baseline and a score of ⩽7 on the GRID-HAMD
  * Week 0 Baseline = Initial baseline assessment
  * Week 5 Waitlist-Period (Delayed Group Only) = 5 weeks post enrollment, but pre-study drug in the Delayed Treatment group only.
  * Week 8 Waitlist-Period (Delayed Group Only) = 8 weeks post enrollment, but pre-study drug in the Delayed Treatment group only.
  * Week 1 Post Psilocybin Treatment = 1 week after the second psilocybin session in both the Immediate Treatment group (Week 5) and Delayed Treatment group (Week 13)
Time Frame: Baseline (Week 0) to 1-week after second psilocybin session (Week 8 in Immediate Treatment; Week 13 in Delayed Treatment). The first psilocybin session (20 mg/70 kg) and second psilocybin session (30 mg/70 kg) are spaced approximately 1 week apart.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment | Delayed Treatment
Number analyzed (Participants) | 13 | 11
units on a scale
  Baseline | 22.9 (3.6) | 22.5 (4.4)
  Week 5 Waitlist-Period (Delayed Group Only) | NA (NA) — This group did not have a waitlist period | 23.8 (5.4)
  Week 8 Waitlist-Period (Delayed Group Only) | NA (NA) — This group did not have a waitlist period | 23.5 (6.0)
  Week 1 Post Psilocybin Treatment | 8.0 (7.1) | 9.5 (8.3)

ADVERSE EVENTS:
Time Frame: Psilocybin session #1 to 1-week after psilocybin session #2 (3 weeks). Immediate treatment group: Weeks 3-5; delayed treatment group: Weeks 11-13.
Description: At each study visit, participants were asked to report on any adverse events since their last study visit. At the psilocybin Session #1, participants were administered 20 mg/70 kg. At the psilocybin Session #2, participants were administered 30 mg/70 kg. Therefore, adverse events are reported here by session number to indicate the rate of adverse events after each drug administration session. No adverse events related to the study were reported prior to drug administration.
Groups:
- Session #1 Through 1-week Post-session #1 Follow-up: Participants received a moderately high psilocybin dose (20 mg/70 kg) in the first session, and were assessed for adverse events at follow-up visits.
- Session #2 Through 1-week Post-session #2 Follow-up: Participants received a high psilocybin dose (30 mg/70 kg) in the second session, and were assessed for adverse events at follow-up visits.
Arm/Group | Session #1 Through 1-week Post-session #1 Follow-up | Session #2 Through 1-week Post-session #2 Follow-up
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 9/24 | 11/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Session #1 Through 1-week Post-session #1 Follow-up (N=24) | Session #2 Through 1-week Post-session #2 Follow-up (N=24)
Headache (Vascular disorders) | 7 (7) | 7 (7)
Physical discomfort (General disorders) | 1 (1) | 0 (0)
Mild controllable muscle motion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Visual distortion (Eye disorders) | 1 (1) | 2 (2)
Tenseness/soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vivid dreams (General disorders) | 0 (0) | 1 (1)
Altered body sensation (General disorders) | 0 (0) | 1 (1)
Blood pressure event (Vascular disorders) | 1 (2) | 0 (0) — A blood pressure event was defined by systolic blood pressure (SBP) > 170 mmHG or diastolic blood pressure (DBP) > 100 mmHg. In these instances, assessments were repeated every 5 minutes until criteria were no longer exceeded.
Heart rate event (Cardiac disorders) | 2 (7) | 2 (5) — A heart rate event was defined by heart rate (HR) > 110 beats per minute. In these instances, assessments were repeated every 5 minutes until criteria were no longer exceeded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03181529/Prot_SAP_000.pdf